CLINICAL TRIAL: NCT04453631
Title: The Efficacy of Transcranial Direct Current Stimulation Combined With the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders: a Double Blind, Sham Controlled, Randomized Factorial Designed Study for Anxiety Disorders
Brief Title: tDCS and Psychotherapy for the Treatment of Anxiety Disorders
Acronym: tDCSplusUP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Ana Ganho Ávila, Integrated Researcher, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS-UP
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Anxiety Disorders
Keywords: anxiety disorders; tDCS; Unified Protocol; RCT
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- active tDCS + CBT-UP (Experimental): Active tDCS combined with the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders.
  Interventions: Device: active tDCS; Behavioral: CBT-UP
- sham tDCS + CBT-UP (Active Comparator): Sham tDCS (control for active tDCS) combined with the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders.
  Interventions: Device: sham tDCS; Behavioral: CBT-UP
- active tDCS + Psychoeducation (Active Comparator): Active tDCS combined with psychoeducation (control condition for CBT-UP).
  Interventions: Device: active tDCS; Behavioral: Psychoeducation
- sham tDCS + Psychoeducation (Placebo Comparator): Sham tDCS combined with psychoeducation (control conditions for active tDCS and CBT-UP).
  Interventions: Device: sham tDCS; Behavioral: Psychoeducation

INTERVENTIONS:
Device: active tDCS — 26 transcranial direct current stimulation sessions, each lasting 20 minutes, with a current intensity of 2 mA, the cathode placed over the right dorsolateral prefrontal cortex and the anode placed over the left deltoid muscle.
  Other Names: Transcranial Direct Current Stimulation
  Arms: active tDCS + CBT-UP; active tDCS + Psychoeducation
Device: sham tDCS — tDCS is controlled in this intervention: sham mode.
  Arms: sham tDCS + CBT-UP; sham tDCS + Psychoeducation
Behavioral: CBT-UP — 15 psychotherapy sessions (1/week) following the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders developed by Barlow et al. 2018.
  Arms: active tDCS + CBT-UP; sham tDCS + CBT-UP
Behavioral: Psychoeducation — To control for the cognitive-behavioral intervention we will use psychoeducation materials.
  Arms: active tDCS + Psychoeducation; sham tDCS + Psychoeducation

SUMMARY:
The main goal of the study is to test the efficacy of tDCS in combination with the Unified Protocol for transdiagnostic treatment of emotional disorders, to reduce anxiety symptoms in a mixed anxiety disorders sample, as assessed by the Hamilton Anxiety Rating Scale (HARS; Hamilton, 1959).

DETAILED DESCRIPTION:
Participants will be randomly allocated to one of four parallel experimental arms, within a 2X2 factorial design in which two interventions (tDCS and CBT-UP) will be delivered, and assessed according to two levels (e.g., intervention vs. no intervention).

Each study participant will assigned to one factor level. Four intervention groups are defined

1. active tDCS + CBT-UP
2. sham tDCS + CBT-UP
3. active tDCS + Psychoeducation
4. sham tDCS + Psychoeducation

The four arms allow to experimentally control the two active therapeutic interventions: active tDCS and CBT-UP. Sham tDCS is the control for active tDCS and psychoeducation is the control condition for CBT-UP.

The intervention will last for 15 weeks, and all groups will comply with the same intervention structure according to the examination plan established in the protocol:

* week 1-2: 1 CBT-UP session/week
* week 3-4: 5 tDCS sessions and 1 CBT-UP session/week
* week 5-8: 2 tDCS sessions and 1 CBT-UP session/week
* week 9-14: 1 tDCS session and 1 CBT-UP session/week
* week 15: 1 CBT-UP session

The treatment will consist of 26 transcranial direct current stimulation sessions, each lasting 20 minutes, with a current intensity of 2 mA, the cathode placed over the right dorsolateral prefrontal cortex and the anode placed over the left deltoid muscle. tDCS will be combined with cognitive-behavioral therapy, in particular following the unified protocol for transdiagnostic treatment of emotional disorders (Barlow et al. 2018).

Safety:

No serious adverse effects are expected with conventional tDCS protocols in humans (≤40 min, ≤4 mA; conclusions from a meta-analysis observing >33200 sessions, >1000 subjects with repeated sessions; Bikson et al., 2016).

Plans for treatment or care after the subject has ended his/her participation in the trial:

Patients will be recommended and offered the best treatment as evidenced by the trial results. For patients that already completed that intervention further standard psychological/psychiatric treatment will be recommended according to patients' status.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of generalized anxiety disorder, specific phobia, panic disorder, agoraphobia, or social anxiety disorder.
* Willing to participate and to give written informed consent

Exclusion Criteria:

1. Contra-indications to tDCS use:

   * Presence of a cardiac or neurological condition
   * Metallic implants
   * If contact with scalp is not possible
   * Have had a head injury resulting in a loss of consciousness that has required further investigation
   * History of seizures
   * Epilepsy or a history of epilepsy
   * Past adverse effects with non-invasive stimulation treatments
2. Current diagnosis of another psychiatric disorder (except for depression, as long as secondary diagnosis), psychoactive medication or psychological treatment
3. Left-handedness
4. Pregnancy
5. Skin condition on the stimulation target area
6. Recreational drug use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-03 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HARS; Hamilton, 1959) | At week 8th, 15th (middle and end of treatment) and 6 months follow-up
  The mean change in the Hamilton Anxiety Rating Scale (HARS; Hamilton, 1959) score, from baseline. HARS total score ranges from 0 to 56, where higher values indicate higher anxiety symptom's severity.

SECONDARY OUTCOMES:
Response to treatment | At week 8th, 15th (middle and end of treatment) and 6 months follow-up.
  Defined as reduction of total Hamilton Anxiety Rating Scale (HARS; Hamilton, 1959) score by ≥ 50%.
Remission to treatment | At week 8th, 15th (middle and end of treatment) and 6 months follow-up.
  Defined as reduction of total Hamilton Anxiety Rating Scale (HARS; Hamilton, 1959) to scores lower than 18 (indicating mild anxiety severity).
Hamilton Depression Rating Scale (HRSD; Hamilton, 1960) | At week 8th, 15th (middle and end of treatment) and 6 months follow-up.
  The mean change in the Hamilton Depression Rating Scale (HRSD; Hamilton, 1960) score, from baseline. HDRS total score ranges from 0 to 75, where higher values indicate higher depressive symptoms' severity.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Barlow DH, Farchione TJ, Bullis JR, Gallagher MW, Murray-Latin H, Sauer-Zavala S, Bentley KH, Thompson-Hollands J, Conklin LR, Boswell JF, Ametaj A, Carl JR, Boettcher HT, Cassiello-Robbins C. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders Compared With Diagnosis-Specific Protocols for Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):875-884. doi: 10.1001/jamapsychiatry.2017.2164. PMID 28768327